CLINICAL TRIAL: NCT03568682
Title: Improving ART Adherence Through Urban Gardening and Peer Nutritional Counseling in the Dominican Republic
Brief Title: Improving Antiretroviral Therapy Adherence Through Urban Gardening and Nutritional Counseling in the Dominican Republic
Acronym: ProMeSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Universidad Autonoma de Santo Domingo (Unknown); Ministerio de Salud Publica, Dominican Republic (Unknown)
Responsible Party: Principal Investigator, Kathryn Derose, Senior Policy Researcher, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R34MH110325 (NIH)
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: HIV
Keywords: food insecurity; nutrition; treatment adherence
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional counseling + urban gardening (Experimental): Participants in the intervention clinic will receive: 1) nutritional counseling from peer counselors in their clinic (approximately 4-5 sessions administered monthly); 2) training from the Ministry of Agriculture on how to plant and maintain a garden in their home (training workshop and monthly follow-up); and 3) a cooking and nutrition workshop facilitated by project nutritionists once garden produce are available.
  Interventions: Behavioral: Nutritional counseling + urban gardening
- Usual care control (No Intervention): Participants in the control clinic will receive their usual care from the clinic. After 12 month follow-up, they will be offered the opportunity to receive the intervention.

INTERVENTIONS:
Behavioral: Nutritional counseling + urban gardening — Peer nutritional counseling and urban gardens
  Arms: Nutritional counseling + urban gardening

SUMMARY:
This pilot study proposes to develop, implement, and evaluate the feasibility, acceptability and preliminary effectiveness of a culturally appropriate, multi-component intervention combining peer nutrition counseling with sustainable urban gardening among people with HIV in the Dominican Republic. The overall hypothesis is that this combined intervention will improve adherence to antiretroviral therapy (ART) and virologic suppression among food insecure HIV+ individuals with suboptimal adherence.

DETAILED DESCRIPTION:
The purpose of this pilot clinical trial is to evaluate the feasibility, acceptability, and preliminary effectiveness of a culturally appropriate, multi-component intervention that targets food insecurity and nutritional health with the ultimate goal of improving antiretroviral therapy adherence and virologic suppression for people with HIV in the Dominican Republic. Through an initial phase, we conducted formative research on dietary patterns and locally available foods and, together with our preliminary research on nutritional counseling and urban gardening, developed a multi-component nutrition intervention to address food insecurity among people with HIV that integrates culturally-appropriate, peer-led nutritional education with a sustainable urban garden component. During the clinical trial phase, we will enroll 120 HIV+ adults with food insecurity and suboptimal adherence in 2 HIV clinics (60 participants in the intervention clinic and 60 participants in the control clinic) and will evaluate the feasibility, acceptability and preliminary effectiveness of urban gardening plus peer nutritional counseling on improving virologic suppression and ART adherence in both the short (month 6) and longer terms (month 12). We will also explore preliminary intervention effects on potential mediators (food security, nutritional status, internalized HIV stigma, and social support). As one of the first studies to develop a sustainable food production approach with peer nutrition counseling among people with HIV, key products will include: 1) an easy-to-use peer nutritional counseling curriculum and urban gardens training materials; 2) pilot data on the feasibility, acceptability, and effects of our intervention on primary outcomes and potential mediators; and 3) if results are promising, an R01 application to conduct a fully-powered cluster randomized controlled trial that examines effects across a larger number of clinics in the Dominican Republic.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ and on ART
* Has moderate or severe household food insecurity
* Has detectable viral load (>50 copies) and/or suboptimal adherence to ART

Exclusion Criteria:

* Does not meet above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in viral load | Change in viral load between baseline and months 6 and 12
  Change in viral load

SECONDARY OUTCOMES:
Antiretroviral therapy adherence | Months 6 and 12
  Self-reported adherence and verified through pharmacy records
HIV care retention | Months 6 and 12
  Self-reported missed clinic visits verified through clinic records

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn P Derose, PhD, MPH, Principal Investigator — RAND
Locations (2):
- Dominican Republic (2):
  - Hospital Regional Dr. Luis Manuel Morillo King, Concepción de la Vega, La Vega
  - Hospital Regional Luis L. Bogaert, Mao, Valverde Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derose KP, Then-Paulino A, Han B, Armenta G, Palar K, Jimenez-Paulino G, Sheira LA, Acevedo R, Fulcar MA, Lugo Bernard C, Veloz Camacho I, Donastorg Y, Wagner GJ. Preliminary Effects of an Urban Gardens and Peer Nutritional Counseling Intervention on HIV Treatment Adherence and Detectable Viral Load Among People with HIV and Food Insecurity: Evidence from a Pilot Cluster Randomized Controlled Trial in the Dominican Republic. AIDS Behav. 2023 Mar;27(3):864-874. doi: 10.1007/s10461-022-03821-3. Epub 2022 Sep 6. PMID 36066760